CLINICAL TRIAL: NCT04237467
Title: Novel Evaluations of Aging and Gender-Affirming Hormone Therapy on Vascular Endothelial Function and Metabolic Profiles in Transgender Men Compared to Age Group-Matched Transgender Women and Cisgender Adults
Brief Title: Effects of Aging and Gender-Affirming Hormone Therapy on Vascular Endothelial Function and Metabolic Profiles in Transgender Men
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-2323
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Transgender; Gender Identity; Vascular Stiffness; Vascular Inflammation; Blood Pressure; Lipid Disorder; Appetitive Behavior
MeSH Terms: conditions — Lipid Metabolism Disorders; Appetitive Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Endothelial cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Older transgender men: This cohort will consist of transgender men aged 50-75 years old who have taken testosterone for at least one year.
  Interventions: Other: No intervention
- Younger transgender men: This cohort will consist of transgender men aged 18-40 years old who have taken testosterone for at least one year.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There was no intervention.

SUMMARY:
This study will examine markers of vascular endothelial function (vascular health) and metabolic profiles in older versus younger transgender men (people who were assigned female at birth but whose gender identity is male). Data will also be compared to those from age group-matched transgender women and cisgender women and men.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-40 years old or 50-75 years old
* Identify as a transgender woman
* Have taken testosterone for at least one year
* Currently taking testosterone parenterally (injections) or transdermally (patches or gels)

Exclusion Criteria:

* Don't identify as a transgender man
* Not currently taking testosterone
* Have been on testosterone for less than one year
* History of hysterectomy/oophorectomy
* Current tobacco smoker
* Current illicit drug use
* History of prior or active estrogen-dependent neoplasms
* Acute liver or gallbladder disease
* Venous thromboembolism
* Hypertriglyceridemia >500 mg/dL
* Fasted plasma glucose >7.0 mmol/L or previously treated diabetes
* Resting blood pressure >140/90 mmHg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender men (people who were assigned female at birth but whose gender identity is male). They may or may not have legally changed their gender marker.
Study Population: Transgender men from the Denver metropolitan area and/or who utilize health care at University of Colorado Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of endothelial function (flow-mediated dilation (FMD) | Baseline
  Brachial artery flow-mediated dilation (FMD), as measured by ultrasound.

SECONDARY OUTCOMES:
Evaluation of carotid artery compliance | Baseline
  The carotid artery compliance index indicates how elastic the artery is. The index describes the change in arterial blood volume in response to a change in arterial blood pressure. Lower numbers are associated with worse outcomes (less elastic arteries).
Evaluation of carotid artery beta stiffness index | Baseline
  The carotid artery beta stiffness index indicates how stiff the artery is. Higher numbers are associated with worse outcomes (stiffer artery)
Carotid artery intimal-medial thickness | Baseline
Evaluation of oxidant burden: oxidized LDL | Baseline
  Oxidized low-density lipoprotein (LDL) measured in the blood and endothelial cells.
Evaluation of oxidant burden: nitrotyrosine | Baseline
  Nitrotyrosine measured in the blood and endothelial cells.
Evaluation of vascular endothelial cell inflammation: NFkB | Baseline
  Protein NFkB (nuclear factor kappa-light-chain-enhancer of activated B cells) measured in blood and endothelial cells.
Evaluation of vascular endothelial cell inflammation: MCP-1 | Baseline
  Monocyte Chemoattractant Protein-1 (MCP-1) measured in blood and endothelial cells.
Evaluation of vascular endothelial cell inflammation: IL-6 | Baseline
  Interleukin 6 (IL-6) measured in blood and endothelial cells.
Evaluation of vascular endothelial cell inflammation: CRP | Baseline
  C-reactive protein (CRP) measured in blood and endothelial cells.
Blood pressure | Baseline
Plasma lipid concentrations: total cholesterol | Baseline
  Total cholesterol will be determined at baseline.
Plasma lipid concentrations: triglycerides | Baseline
  Triglycerides will be determined at baseline.
Insulin sensitivity | Baseline
Whole body composition: Percent Lean Mass | Baseline
  Percent lean mass will be determined using dual energy x-ray absorptiometry.
Whole body composition: Percent Fat Mass | Baseline
  Percent fat mass will be determined using dual energy x-ray absorptiometry.
Regional body composition: Percent Lean Mass | Baseline
  Regional percent lean mass will be determined using dual energy x-ray absorptiometry.
Regional body composition: Percent Fat Mass | Baseline
  Regional percent fat mass will be determined using dual energy x-ray absorptiometry.
Body weight | Baseline
Appetite ratings | Baseline
Appetite-related peptides | Baseline
D-Dimer | Baseline
Alcohol use | Baseline
Depression symptoms | Baseline
Physical activity monitoring | 7 days
  Physical activity will me monitored for 7 days with an ActivPALmonitor
Energy intake | 3 days
  Energy intake will be estimated with a 3-day food diary

CONTACTS AND LOCATIONS:
Overall Officials: Sean Iwamoto, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No